CLINICAL TRIAL: NCT01930487
Title: The Effects of an Antioxidant Formulation on Intraocular Pressure, Ocular Perfusion Pressure, Retrobulbar, Retinal Capillary and Choroidal Blood Flow
Brief Title: The Effects of an Antioxidant Formulation on Ocular Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ScienceBased Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 007
Record Dates: First submitted 2013-08-09; First posted 2013-08-29 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-01

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Primary open angle glaucoma; intraocular pressure; ocular perfusion pressure; retrobulbar blood flow; retinal capillary blood flow; choroidal blood flow
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Dietary Supplements; Antioxidants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- supplement w/ antioxidants then placebo (Experimental): dietary supplement with antioxidants, followed by placebo supplement
  Interventions: Dietary Supplement: dietary supplement with antioxidants; Dietary Supplement: Placebo
- placebo then supplement w/ antioxidants (Experimental): placebo supplement, followed by dietary supplement with antioxidants
  Interventions: Dietary Supplement: dietary supplement with antioxidants; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: dietary supplement with antioxidants — Formulation contains vitamins, a mineral, dietary antioxidants, amino acids, polyphenols and polyunsaturated fatty acids
  Other Names: Optic Nerve Formula
Dietary Supplement: Placebo — Placebo - Softgels manufactured to mimic the appearance of active, dietary supplement with antioxidants

SUMMARY:
The objective is to evaluate the effects of an antioxidant formula versus placebo on ocular blood flow in a randomized double-blind, crossover design.

Based upon preliminary data, it is hypothesized that a dietary supplement containing a variety of ingredients with antioxidant properties will, compared to placebo, increase ocular perfusion pressure, retrobulbar, retinal capillary and choroidal blood flow, and maintain these effects over the course of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 years or older.
* Confirmed diagnosis of open angle glaucoma by glaucoma specialist in the study eye, as evidenced from criteria representative of glaucomatous optic nerve damage such as specific optic disc or retinal nerve fiber layer structural abnormalities and/or visual field abnormalities.
* Best corrected visual acuity at 20/60 or better in study eye.
* Willingness to avoid caffeine and smoking for 12 hours before and during the study visits.

Exclusion Criteria:

* History of acute angle-closure or a narrow, occluding of anterior chamber angle by gonioscopy.
* History of chronic or recurrent inflammatory eye diseases or signs of intraocular trauma and/or unreliable applanation tonometry.
* Severe, unstable or uncontrolled cardiovascular, renal or pulmonary disease
* History of/or current renal or hepatic impairment.
* History of/or current bronchial asthma, severe chronic obstructive pulmonary disease, sinus bradycardia, second or third degree atrioventricular block, or cardiogenic shock.
* Recent surgery or surgery planned near study timeline
* History of bleeding disorder
* Use of blood thinning medications
* Use of specified dietary supplements for three weeks prior to study entry and throughout study period.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-08; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alon Harris, PhD, Principal Investigator — Professor of Ophthalmology, Professor of Cellular and Integrative Physiology, Director Clinical Research Glick Eye Institute, Indiana University Medical Center
Locations (1):
- Glick Eye Institute, Ocular Vascular Research Center, Indiana University School of Medicine, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 47 patients were recruited for the study
Pre-assignment Details: 1 subject started but did not complete the baseline examination and was not randomized to either treatment arm.
Groups:
- Supplement With Antioxidants, Then Placebo: dietary supplement with antioxidants in the first intervention period, followed by placebo supplement in the second intervention period
- Placebo, Then Supplement With Antioxidants: placebo supplement in the second intervention period, followed by dietary supplement with antioxidants in the second intervention period
Period: First Intervention (30 Days)
Arm/Group | Supplement With Antioxidants, Then Placebo | Placebo, Then Supplement With Antioxidants
Started | 21 | 25
Completed | 19 | 23
Not Completed | 2 | 2
Period: Washout Period (3 Weeks)
Arm/Group | Supplement With Antioxidants, Then Placebo | Placebo, Then Supplement With Antioxidants
Started | 19 | 23
Completed | 19 | 23
Not Completed | 0 | 0
Period: Second Intervention (30 Days)
Arm/Group | Supplement With Antioxidants, Then Placebo | Placebo, Then Supplement With Antioxidants
Started | 19 | 23
Completed | 19 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: patients who completed both periods of the crossover study
Groups:
- Participants Completing Study: Participants who completed both arms of the crossover study
Arm/Group | Participants Completing Study
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 34
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 42
Diabetes (Type 2) [Number; unit: participants]
  yes | 21
  no | 21
Hypertension [Number; unit: participants]
  yes | 16
  no | 26
Study Eye [Number; unit: participants]
  right | 24
  left | 18
Duration of OAG [Mean (Standard Deviation); unit: years] | 15 (8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Superior Retinal Capillary Blood Flow (% Zero Pixels)
Description: change (post-treatment - pre-treatment) in superior retinal capillary blood flow (% zero pixels or % avascular tissue) using Heidelberg Retinal Flowmeter (HRF)
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: % zero pixels
Groups:
- Dietary Supplement With Antioxidants: Dietary supplement with antioxidants, Ginkgo biloba, Bilberry extract
  dietary supplement with antioxidants: Formulation contains vitamins, a mineral, dietary antioxidants, amino acids, polyphenols and polyunsaturated fatty acids
- Placebo: Placebo identical in appearance to active
  Softgels manufactured to mimic the appearance of active dietary supplement with antioxidants
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 42 | 42
% zero pixels | -0.026 (0.008) | 0.011 (0.007)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0016, paired t-test, 2-sided; Mean Difference (Net) = -0.037, Standard Error of Mean 0.011 — dietary supplement with antioxidants - placebo

2. Primary Outcome: Change in Inferior Retinal Capillary Blood Flow (% Zero Pixels)
Description: change (post-treatment - pre-treatment) in inferior retinal capillary blood flow (% zero pixels or % avascular tissue) using Heidelberg Retinal Flowmeter (HRF)
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: % zero pixels
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 42 | 42
% zero pixels | -0.016 (0.007) | 0.009 (0.007)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0249, paired t-test, 2-sided; Mean Difference (Net) = -0.025, Standard Error of Mean 0.011 — dietary supplement with antioxidants - placebo

3. Secondary Outcome: Change in Ocular Perfusion Pressure
Description: change (post-treatment - pre-treatment) in ocular perfusion pressure (2/3 Mean arterial pressure - intraocular pressure)
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 42 | 42
mm Hg | 1.5 (0.9) | 1.4 (1.2)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.9147, paired t-test, 2-sided; Mean Difference (Net) = 0.1, Standard Error of Mean 1.3 — dietary supplement with antioxidants - placebo

4. Secondary Outcome: Change in Ophthalmic Artery Peak Systolic Blood Flow Velocity (cm/s)
Description: change (post-treatment - pre-treatment) in ophthalmic artery peak systolic blood flow velocity (cm/s) using color Doppler imaging (CDI)
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 42 | 42
cm/s | 0.74 (0.41) | -0.94 (0.38)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0070, paired t-test, 2-sided; Mean Difference (Net) = 1.67, Standard Error of Mean 0.59 — dietary supplement with antioxidants - placebo

5. Secondary Outcome: Change in Central Retinal Artery Peak Systolic Blood Flow Velocity (cm/s)
Description: change (post-treatment - pre-treatment) in central retinal artery peak systolic blood flow velocity (cm/s) using color Doppler imaging (CDI)
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 42 | 42
cm/s | 0.54 (0.15) | -0.43 (0.15)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p < 0.0001, paired t-test, 2-sidede; Mean Difference (Net) = 0.97, Standard Error of Mean 0.21 — dietary supplement with antioxidants - placebo

6. Secondary Outcome: Change in Nasal Posterior Ciliary Artery Peak Systolic Blood Flow Velocity (cm/s)
Description: change (post-treatment - pre-treatment) in nasal posterior ciliary artery peak systolic blood flow velocity (cm/s) using color Doppler imaging (CDI)
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 42 | 42
cm/s | 0.30 (0.14) | -0.16 (0.16)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0476, paired t-test, 2-sided; Mean Difference (Net) = 0.46, Standard Error of Mean 0.23 — dietary supplement with antioxidants - placebo

7. Secondary Outcome: Change in Temporal Posterior Ciliary Artery Peak Systolic Blood Flow Velocity (cm/s)
Description: change (post-treatment - pre-treatment) in temporal posterior ciliary artery peak systolic blood flow velocity (cm/s) using color Doppler imaging (CDI)
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 42 | 42
cm/s | 0.31 (0.16) | -0.14 (0.15)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0352, paired t-test, 2-sided; Mean Difference (Net) = 0.45, Standard Error of Mean 0.21 — dietary supplement with antioxidants - placebo

8. Secondary Outcome: Change in Ophthalmic Artery End Diastolic Blood Flow Velocity (cm/s)
Description: change (post-treatment - pre-treatment) in ophthalmic artery end diastolic blood flow velocity (cm/s) using color Doppler imaging (CDI)
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 42 | 42
cm/s | 0.35 (0.13) | -0.17 (0.17)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0208, paired t-test, 2-sided; Mean Difference (Net) = 0.51, Standard Error of Mean 0.21 — dietary supplement with antioxidants - placebo

9. Secondary Outcome: Change in Central Retinal Artery End Diastolic Blood Flow Velocity (cm/s)
Description: change (post-treatment - pre-treatment) in central retinal artery end diastolic blood flow velocity (cm/s) using color Doppler imaging (CDI)
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 42 | 42
cm/s | 0.27 (0.05) | -0.11 (0.06)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p < 0.0001, paired t-test, 2-sided; Mean Difference (Net) = 0.38, Standard Error of Mean 0.07 — dietary supplement with antioxidants - placebo

10. Secondary Outcome: Change in Nasal Posterior Ciliary Artery End Diastolic Blood Flow Velocity (cm/s)
Description: change (post-treatment - pre-treatment) in nasal posterior ciliary artery end diastolic blood flow velocity (cm/s) using color Doppler imaging (CDI)
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 42 | 42
cm/s | 0.17 (0.05) | -0.07 (0.05)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0024, paired t-test, 2-sided; Mean Difference (Net) = 0.24, Standard Error of Mean 0.07 — dietary supplement with antioxidants - placebo

11. Secondary Outcome: Change in Temporal Posterior Ciliary Artery End Diastolic Blood Flow Velocity (cm/s)
Description: change (post-treatment - pre-treatment) in temporal posterior ciliary artery end diastolic blood flow velocity (cm/s) using color Doppler imaging (CDI)
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 42 | 42
cm/s | 0.15 (0.05) | -0.06 (0.05)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0081, paired t-test, 2-sided; Mean Difference (Net) = 0.21, Standard Error of Mean 0.07 — dietary supplement with antioxidants - placebo

12. Secondary Outcome: Change in Ophthalmic Artery Blood Flow - Vascular Resistance (Ratio)
Description: change (post-treatment - pre-treatment) in ophthalmic artery blood flow - vascular resistance (ratio) using color Doppler imaging (CDI)
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 42 | 42
ratio | -0.007 (0.004) | -0.005 (0.006)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.8191, paired t-test, 2-sided; Mean Difference (Net) = -0.002, Standard Error of Mean 0.008 — dietary supplement with antioxidants - placebo

13. Secondary Outcome: Change in Central Retinal Artery Blood Flow - Vascular Resistance (Ratio)
Description: change (post-treatment - pre-treatment) in central retinal artery blood flow - vascular resistance (ratio) using color Doppler imaging (CDI)
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 42 | 42
ratio | -0.018 (0.006) | 0.000 (0.006)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0482, paired t-test, 2-sided; Mean Difference (Net) = -0.018, Standard Error of Mean 0.009 — dietary supplement with antioxidants - placebo

14. Secondary Outcome: Change in Nasal Posterior Ciliary Artery Blood Flow - Vascular Resistance (Ratio)
Description: change (post-treatment - pre-treatment) in nasal posterior ciliary artery blood flow - vascular resistance (ratio) using color Doppler imaging (CDI)
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 42 | 42
ratio | -0.013 (0.006) | 0.005 (0.005)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0230, paired t-test, 2-sided; Mean Difference (Net) = -0.019, Standard Error of Mean 0.0230 — dietary supplement with antioxidants - placebo

15. Secondary Outcome: Change in Temporal Posterior Ciliary Artery Blood Flow - Vascular Resistance (Ratio)
Description: change (post-treatment - pre-treatment) in temporal posterior ciliary artery blood flow - vascular resistance (ratio) using color Doppler imaging (CDI)
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 42 | 42
ratio | -0.009 (0.006) | 0.004 (0.005)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.1202, paired t-test, 2-sided; Mean Difference (Net) = -0.013, Standard Error of Mean 0.008 — dietary supplement with antioxidants - placebo

16. Secondary Outcome: Change in Ophthalmic Artery Peak Systolic Blood Flow Velocity (cm/s) - DM
Description: change (post-treatment - pre-treatment) in ophthalmic artery peak systolic blood flow velocity (cm/s) using color Doppler imaging (CDI) in patients with type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
cm/s | 1.71 (0.56) | -0.84 (0.48)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0063, paired t-test, 2-sided; Mean Difference (Net) = 2.55, Standard Error of Mean 0.83 — dietary supplement with antioxidants - placebo

17. Secondary Outcome: Change in Ophthalmic Artery Peak Systolic Blood Flow Velocity (cm/s) - No DM
Description: change (post-treatment - pre-treatment) in ophthalmic artery peak systolic blood flow velocity (cm/s) using color Doppler imaging (CDI) in patients without type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
cm/s | -0.24 (0.53) | -1.03 (0.60)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.3347, paired t-test, 2-sided; Mean Difference (Net) = 0.80, Standard Error of Mean 0.80 — dietary supplement with antioxidants - placebo

18. Secondary Outcome: Change in Central Retinal Artery Peak Systolic Blood Flow Velocity (cm/s) - DM
Description: change (post-treatment - pre-treatment) in central retinal artery peak systolic blood flow velocity (cm/s) using color Doppler imaging (CDI) in patients with type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
cm/s | 0.58 (0.20) | -0.44 (0.24)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0094, paired t-test, 2-sided; Mean Difference (Net) = 1.02, Standard Error of Mean 0.35 — dietary supplement with antioxidants - placebo

19. Secondary Outcome: Change in Central Retinal Artery Peak Systolic Blood Flow Velocity (cm/s) - No DM
Description: change (post-treatment - pre-treatment) in central retinal artery peak systolic blood flow velocity (cm/s) using color Doppler imaging (CDI) in patients without type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
cm/s | 0.51 (0.23) | -0.41 (0.20)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0009, paired t-test, 2-sided; Mean Difference (Net) = 0.92, Standard Error of Mean 0.24 — dietary supplement with antioxidants - placebo

20. Secondary Outcome: Change in Nasal Posterior Ciliary Artery Peak Systolic Blood Flow Velocity (cm/s) - DM
Description: change (post-treatment - pre-treatment) in nasal posterior ciliary artery peak systolic blood flow velocity (cm/s) using color Doppler imaging (CDI) in patients with type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
cm/s | 0.56 (0.22) | -0.46 (0.23)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0067, paired t-test, 2-sided; Mean Difference (Net) = 1.02, Standard Error of Mean 0.34 — dietary supplement with antioxidants - placebo

21. Secondary Outcome: Change in Nasal Posterior Ciliary Artery Peak Systolic Blood Flow Velocity (cm/s) - No DM
Description: change (post-treatment - pre-treatment) in nasal posterior ciliary artery peak systolic blood flow velocity (cm/s) using color Doppler imaging (CDI) in patients without type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
cm/s | 0.03 (0.16) | 0.13 (0.22)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.6938, paired t-test, 2-sided; Mean Difference (Net) = -0.10, Standard Error of Mean 0.25 — dietary supplement with antioxidants - placebo

22. Secondary Outcome: Change in Temporal Posterior Ciliary Artery Peak Systolic Blood Flow Velocity (cm/s) - DM
Description: change (post-treatment - pre-treatment) in temporal posterior ciliary artery peak systolic blood flow velocity (cm/s) using color Doppler imaging (CDI) in patients with type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
cm/s | 0.24 (0.19) | -0.32 (0.21)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0805, paired t-test, 2-sided; Mean Difference (Net) = 0.56, Standard Error of Mean 0.30 — dietary supplement with antioxidants - placebo

23. Secondary Outcome: Change in Temporal Posterior Ciliary Artery Peak Systolic Blood Flow Velocity (cm/s) - No DM
Description: change (post-treatment - pre-treatment) in temporal posterior ciliary artery peak systolic blood flow velocity (cm/s) using color Doppler imaging (CDI) in patients without type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
cm/s | 0.38 (0.27) | 0.03 (0.21)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.2451, paired t-test, 2-sided; Mean Difference (Net) = 0.35, Standard Error of Mean 0.29 — dietary supplement with antioxidants - placebo

24. Secondary Outcome: Change in Ophthalmic Artery End Diastolic Blood Flow Velocity (cm/s) - DM
Description: change (post-treatment - pre-treatment) in ophthalmic artery end diastolic blood flow velocity (cm/s) using color Doppler imaging (CDI) in patients with type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
cm/s | 0.60 (0.19) | -0.18 (0.24)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0323, paired t-test, 2-sided; Mean Difference (Net) = 0.78, Standard Error of Mean 0.34 — dietary supplement with antioxidants - placebo

25. Secondary Outcome: Change in Ophthalmic Artery End Diastolic Blood Flow Velocity (cm/s) - No DM
Description: change (post-treatment - pre-treatment) in ophthalmic artery end diastolic blood flow velocity (cm/s) using color Doppler imaging (CDI) in patients without type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
cm/s | 0.09 (0.18) | -0.16 (0.24)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.3440, paired t-test, 2-sided; Mean Difference (Net) = 0.25, Standard Error of Mean 0.26 — dietary supplement with antioxidants - placebo

26. Secondary Outcome: Change in Central Retinal Artery End Diastolic Blood Flow Velocity (cm/s) - DM
Description: change (post-treatment - pre-treatment) in central retinal artery end diastolic blood flow velocity (cm/s) using color Doppler imaging (CDI) in patients with type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
cm/s | 0.29 (0.06) | -0.08 (0.11)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0119, paired t-test, 2-sided; Mean Difference (Net) = 0.37, Standard Error of Mean 0.13 — dietary supplement with antioxidants - placebo

27. Secondary Outcome: Change in Central Retinal Artery End Diastolic Blood Flow Velocity (cm/s) - No DM
Description: change (post-treatment - pre-treatment) in central retinal artery end diastolic blood flow velocity (cm/s) using color Doppler imaging (CDI) in patients without type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
cm/s | 0.26 (0.07) | -0.14 (0.07)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p < 0.0001, paired t-test, 2-sided; Mean Difference (Net) = 0.40, Standard Error of Mean 0.07 — dietary supplement with antioxidants - placebo

28. Secondary Outcome: Change in Nasal Posterior Ciliary Artery End Diastolic Blood Flow Velocity (cm/s) - DM
Description: change (post-treatment - pre-treatment) in nasal posterior ciliary artery end diastolic blood flow velocity (cm/s) using color Doppler imaging (CDI) in patients with type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
cm/s | 0.16 (0.07) | -0.16 (0.08)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0137, paired t-test, 2-sided; Mean Difference (Net) = 0.32, Standard Error of Mean 0.12 — dietary supplement with antioxidants - placebo

29. Secondary Outcome: Change in Nasal Posterior Ciliary Artery End Diastolic Blood Flow Velocity (cm/s) - No DM
Description: change (post-treatment - pre-treatment) in nasal posterior ciliary artery end diastolic blood flow velocity (cm/s) using color Doppler imaging (CDI) in patients without type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
cm/s | 0.18 (0.07) | 0.01 (0.07)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0866, paired t-test, 2-sided; Mean Difference (Net) = 0.16, Standard Error of Mean 0.09 — dietary supplement with antioxidants - placebo

30. Secondary Outcome: Change in Temporal Posterior Ciliary Artery End Diastolic Blood Flow Velocity (cm/s) - DM
Description: change (post-treatment - pre-treatment) in temporal posterior ciliary artery end diastolic blood flow velocity (cm/s) using color Doppler imaging (CDI) in patients with type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
cm/s | 0.10 (0.07) | -0.13 (0.07)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0656, paired t-test, 2-sided; Mean Difference (Net) = 0.23, Standard Error of Mean 0.12 — dietary supplement with antioxidants - placebo

31. Secondary Outcome: Change in Temporal Posterior Ciliary Artery End Diastolic Blood Flow Velocity (cm/s) - No DM
Description: change (post-treatment - pre-treatment) in temporal posterior ciliary artery end diastolic blood flow velocity (cm/s) using color Doppler imaging (CDI) in patients without type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: cm/s
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
cm/s | 0.20 (0.08) | 0.01 (0.08)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0626, paired t-test, 2-sided; Mean Difference (Net) = 0.19, Standard Error of Mean 0.09 — dietary supplement with antioxidants - placebo

32. Secondary Outcome: Change in Ophthalmic Artery Blood Flow - Vascular Resistance (Ratio) - DM
Description: change (post-treatment - pre-treatment) in ophthalmic artery blood flow - vascular resistance (ratio) using color Doppler imaging (CDI) in patients with type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
ratio | -0.008 (0.007) | -0.005 (0.009)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.8100, paired t-test, 2-sided; Mean Difference (Net) = -0.003, Standard Error of Mean 0.013 — dietary supplement with antioxidants - placebo

33. Secondary Outcome: Change in Ophthalmic Artery Blood Flow - Vascular Resistance (Ratio) - No DM
Description: change (post-treatment - pre-treatment) in ophthalmic artery blood flow - vascular resistance (ratio) using color Doppler imaging (CDI) in patients without type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
ratio | -0.005 (0.006) | -0.004 (0.009)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.9556, paired t-test, 2-sided; Mean Difference (Net) = -0.001, Standard Error of Mean 0.010 — dietary supplement with antioxidants - placebo

34. Secondary Outcome: Change in Central Retinal Artery Blood Flow - Vascular Resistance (Ratio) - DM
Description: change (post-treatment - pre-treatment) in central retinal artery blood flow - vascular resistance (ratio) using color Doppler imaging (CDI) in patients with type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
ratio | -0.019 (0.010) | -0.004 (0.011)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.3414, paired t-test, 2-sided; Mean Difference (Net) = -0.015, Standard Error of Mean 0.015 — dietary supplement with antioxidants - placebo

35. Secondary Outcome: Change in Central Retinal Artery Blood Flow - Vascular Resistance (Ratio) - No DM
Description: change (post-treatment - pre-treatment) in central retinal artery blood flow - vascular resistance (ratio) using color Doppler imaging (CDI) in patients without type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
ratio | -0.017 (0.007) | 0.004 (0.007)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0330, paired t-test, 2-sided; Mean Difference (Net) = -0.021, Standard Error of Mean 0.009 — dietary supplement with antioxidants - placebo

36. Secondary Outcome: Change in Nasal Posterior Artery Blood Flow - Vascular Resistance (Ratio) - DM
Description: change (post-treatment - pre-treatment) in nasal posterior artery blood flow - vascular resistance (ratio) using color Doppler imaging (CDI) in patients with type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
ratio | -0.005 (0.007) | 0.005 (0.007)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.3326, paired t-test, 2-sided; Mean Difference (Net) = -0.010, Standard Error of Mean 0.010 — dietary supplement with antioxidants - placebo

37. Secondary Outcome: Change in Nasal Posterior Artery Blood Flow - Vascular Resistance (Ratio) - No DM
Description: change (post-treatment - pre-treatment) in nasal posterior artery blood flow - vascular resistance (ratio) using color Doppler imaging (CDI) in patients without type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
ratio | -0.022 (0.010) | 0.005 (0.007)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0348, paired t-test, 2-sided; Mean Difference (Net) = -0.027, Standard Error of Mean 0.012 — dietary supplement with antioxidants - placebo

38. Secondary Outcome: Change in Temporal Posterior Artery Blood Flow - Vascular Resistance (Ratio) - DM
Description: change (post-treatment - pre-treatment) in temporal posterior artery blood flow - vascular resistance (ratio) using color Doppler imaging (CDI) in patients with type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
ratio | -0.006 (0.009) | 0.010 (0.007)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.2089, paired t-test, 2-sided; Mean Difference (Net) = -0.016, Standard Error of Mean 0.012 — dietary supplement with antioxidants - placebo

39. Secondary Outcome: Change in Temporal Posterior Artery Blood Flow - Vascular Resistance (Ratio) - No DM
Description: change (post-treatment - pre-treatment) in temporal posterior artery blood flow - vascular resistance (ratio) using color Doppler imaging (CDI) in patients without type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
ratio | -0.012 (0.009) | -0.001 (0.007)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.3738, paired t-test, 2-sided; Mean Difference (Net) = -0.010, Standard Error of Mean 0.012 — dietary supplement with antioxidants - placebo

40. Secondary Outcome: Change in Ocular Perfusion Pressure - DM
Description: change (post-treatment - pre-treatment) in Ocular perfusion pressure in patients with type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
mm Hg | 0.2 (1.2) | -1.1 (1.4)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.4470, paired t-test, 2-sided; Mean Difference (Net) = 1.3, Standard Error of Mean 1.7 — dietary supplement with antioxidants - placebo

41. Secondary Outcome: Change in Ocular Perfusion Pressure - No DM
Description: change (post-treatment - pre-treatment) in Ocular perfusion pressure in patients without type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
mm Hg | 2.8 (1.4) | 3.8 (1.7)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.6382, paired t-test, 2-sided; Mean Difference (Net) = -1.0, Standard Error of Mean 2.1 — dietary supplement with antioxidants - placebo

42. Secondary Outcome: Change in Superior Retinal Capillary Blood Flow (% Zero Pixels) - DM
Description: change (post-treatment - pre-treatment) in superior retinal capillary blood flow (% zero pixels or % avascular tissue) using Heidelberg Retinal Flowmeter (HRF) in patients with type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: % zero pixels
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
% zero pixels | -0.031 (0.009) | 0.012 (0.010)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0026, paird t-test, 2-sided; Mean Difference (Net) = -0.043, Standard Error of Mean 0.012 — dietary supplement with antioxidants - placebo

43. Secondary Outcome: Change in Superior Retinal Capillary Blood Flow (% Zero Pixels) - No DM
Description: change (post-treatment - pre-treatment) in superior retinal capillary blood flow (% zero pixels or % avascular tissue) using Heidelberg Retinal Flowmeter (HRF) in patients without type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: % zero pixels
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
% zero pixels | -0.021 (0.014) | 0.010 (0.009)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.1045, paired t-test, 2-sided; Mean Difference (Net) = -0.030, Standard Error of Mean 0.018 — dietary supplement with antioxidants - placebo

44. Secondary Outcome: Change in Inferior Retinal Capillary Blood Flow (% Zero Pixels) - DM
Description: change (post-treatment - pre-treatment) in inferior retinal capillary blood flow (% zero pixels or % avascular tissue) using Heidelberg Retinal Flowmeter (HRF) in patients with type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: % zero pixels
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
% zero pixels | -0.005 (0.009) | 0.000 (0.008)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.6941, paired t-test; Mean Difference (Net) = -0.005, Standard Error of Mean 0.013 — dietary supplement with antioxidants - placebo

45. Secondary Outcome: Change in Inferior Retinal Capillary Blood Flow (% Zero Pixels) - No DM
Description: change (post-treatment - pre-treatment) in inferior retinal capillary blood flow (% zero pixels or % avascular tissue) using Heidelberg Retinal Flowmeter (HRF) in patients without type 2 diabetes
Time Frame: baseline and 30 days
Population: patients completing both study periods
Measure: Mean (Standard Error); unit: % zero pixels
Arm/Group | Dietary Supplement With Antioxidants | Placebo
Number analyzed (Participants) | 21 | 21
% zero pixels | -0.028 (0.009) | 0.018 (0.010)
Statistical Analysis 1: Comparison: Dietary Supplement With Antioxidants vs Placebo; Test type: Superiority or Other; p = 0.0138, paired t-test, 2-sided; Mean Difference (Net) = -0.046, Standard Error of Mean 0.017 — dietary supplement with antioxidants - placebo

ADVERSE EVENTS:
Time Frame: Four weeks for each intervention, with a 3-week wash out period between interventions
Description: Safety population included all participants who completed study. (45 patients with OAG were enrolled, 42 of which were followed through to completion of the study. Three patients discontinued study participation due to difficulty in adhering to study visit timeline.)
Groups:
- Supplement w/ Antioxidants: dietary supplement with antioxidants
  dietary supplement with antioxidants: Formulation contains vitamins, a mineral, dietary antioxidants, amino acids, polyphenols and polyunsaturated fatty acids
- Placebo: placebo supplement
  Placebo: Placebo - Softgels manufactured to mimic the appearance of active, dietary supplement with antioxidants
Arm/Group | Supplement w/ Antioxidants | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No